CLINICAL TRIAL: NCT06832085
Title: Combination Nicotine Replacement Therapy, Cytisine, or Varenicline for Smoking Cessation: A Randomized Controlled Trial
Brief Title: Combination Nicotine Replacement Therapy, Cytisine, or Varenicline for Smoking Cessation
Acronym: Sun Life RCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Sun Life Assurance Company of Canada (Unknown); Vita Aid Professional Therapeutics (Unknown); Lumino Health™ Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240741-01H
Record Dates: First submitted 2025-01-21; First posted 2025-02-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-01

CONDITIONS: Tobacco
Keywords: Tobacco; Tobacco cessation; Nicotine; Nicotine replacement therapy; Cytisine; Varenicline; counselling
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; cytisine; Varenicline

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nicotine Replacement Therapy (Nicotine patch plus NRT gum or lozenge) (Active Comparator): Nicotine replacement therapy patch (titrated based on cigarettes consumed at baseline) plus short term gum or lozenge (as needed)
  Interventions: Drug: Nicotine Replacement Therapy (Nicotine patch plus NRT gum or lozenge)
- Cytisine (Active Comparator): Cytisine pills, standard dose
  Interventions: Drug: Cytisine
- Varenicline (Champix) (Active Comparator): Varenicline - standard dose
  Interventions: Drug: Varenicline (Champix)

INTERVENTIONS:
Drug: Nicotine Replacement Therapy (Nicotine patch plus NRT gum or lozenge) — Participants in this group will apply 1 NRT patch each morning for up to 26 weeks. Patches will be titrated based on cigarettes consumed. Short-acting NRT products (gum and lozenge) will be used as needed by the participants in this group.
  Other Names: Nicotine Replacement Therapy gum; Nicotine Replacement Therapy lozenge
  Arms: Nicotine Replacement Therapy (Nicotine patch plus NRT gum or lozenge)
Drug: Cytisine — Participants in this group will take 3mg of cytisine 3 times per day for 12 weeks.
  Arms: Cytisine
Drug: Varenicline (Champix) — Participants in this group will take 1mg of varenicline 2 times per day for 12 weeks.
  Arms: Varenicline (Champix)

SUMMARY:
The purpose of this trial is to test whether clients of Sun Life are willing to join in a quit smoking program that offers counselling and tobacco cessation products to all participants over a 12-month period. The study team will track the safety and usage of 3 types of cessation products as well as the effectiveness of a virtual pharmacy (i.e. cessation products delivered to participants directly from a pharmacy) over a 12-week treatment period.

The purpose of this study is to look at 3 approved smoking cessation products used in combination with counselling and virtual delivery of the smoking cessation products. The goal is to track product usage, safety, and adherence (how much of the products people use and how many counselling sessions they complete).

Within the study there will also be an observational group who will not receive study medication but who will receive free virtual coaching and follow-up for smoking cessation and complete study questionnaires.

DETAILED DESCRIPTION:
This study will engage people who smoke through an insurance-based outreach program (Sun Life Assurance Company of Canada) to evaluate the efficacy and safety of three pharmacotherapy arms (combination NRT, cytisine, or varenicline) within the OMSC framework, which includes the provision of cost-free virtual counselling, follow-up, and direct-to-consumer delivery of medications.

To our knowledge, there are no prior studies evaluating an entirely virtual smoking cessation intervention which includes virtual counselling/follow-up and direct-to-consumer delivery of pharmacotherapy. This study will also engage the broader community setting, such as clients or employees of industry partners, represents a valuable opportunity to reach a wider population of people who smoke with tailored support. Beyond cost savings associated with smoking cessation, this study may also reduce insurance premiums for patients, thus leading to additional source of cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Current cigarette smokers (more than 5 cigarettes per day) who are interested in reducing or quitting in the next 6 months.
* Able to provide informed consent.
* Living in Ontario, Canada

Exclusion Criteria:

* Contraindications to any of the study medications (NRT, cytisine, varenicline).
* Actively using one of the study medications in the past 7 days.
* Actively enrolled in another formal smoking cessation program.
* Pregnant or breastfeeding individuals.
* Unable to engage in follow-up for any reason (for example an acute mental illness, cognitive impairment, unable to speak English or French).
* Other conditions deemed by the study team to interfere with participation or outcomes in the opinion of the study investigator (for example acutely unwell, life expectancy less than 1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant's Smoking Status | 6 months
  7-Day Point Prevalence of Smoking Cessation will be measured at 6 months. For those who report they have quit smoking, this will be biochemically verified through a salivary cotinine test.

SECONDARY OUTCOMES:
Participant's Smoking Status at follow-up | 1, 3, and 12 months
  7-Day Point Prevalence of Smoking Cessation will be measured at each follow-up time point via survey. For those who report they have quit smoking, this will be biochemically verified through a salivary cotinine test.
Number of quit attempts made by participant | 6, and 12 months
  Participants will be asked via survey at each follow-up visit if they have had a reduction in their cigarette consumption or made a quit attempt (defined as abstaining from tobacco for at least 24-hours). If they have made a quit attempt, they will be asked to report how many quit attempts they have made since the last follow-up visit. The total number of times the participant has refrained from using tobacco for at least 24-hours will be recorded.
Participant's level of nicotine dependance | 6, and 12 months
  Participants will be asked via survey response to complete the Fagerstrom Test for Nicotine Dependence at each follow-up visit. The total score will be calculated and recorded for each time point.
Participant's heaviness of smoking score | 6, and 12 months
  Participants will be asked via survey response to complete the Heaviness of Smoking Index (to record the current level of dependence) at each follow-up visit. The total score will be calculated and recorded for each time point.
Participant's adherence to the counselling program | 12 months
  Attendance will be recorded for each counselling visit and adherence will be totaled for each participant at the end of the study.
Participant's adherence to study medication | 6 months
  Adherence to the prescribed medication and regime will be collected for each participant via self-report. The number of weeks on treatment will be recorded along with the number of missed doses.
Participant's response to smoking cessation quality of life questionnaire | Baseline, 6 and 12 months
  The tobacco specific SF-36 questionnaire will be administered at each follow-up visit. The total score will be recorded for each visit.
Participant's response to the Patient Health Questionnaire (PHQ-9) | Baseline, 6 and 12 months
  The PHQ-9 will be administered at each follow-up visit. The score will be calculated and recorded for each participant.
Participant's response to the General Anxiety Disorder Questionnaire (GAD-7) | Baseline, 6 and 12 months
  The GAD-7 will be administered at each follow-up visit. The score will be calculated and recorded for each participant.

OTHER OUTCOMES:
Participant recruitment metrics | 12 months
  The number of Sun Life clients emailed and the number of clients who click the link to self-refer to the program will be recorded by Sun Life and reported to the study team at the end of the study. This will be compared to the number of people screened and enrolled by the study team.
Participant satisfaction metrics | 12 months
  At the end of study participation, participants will be asked a series of satisfaction questions related to their counselling sessions (information provided, length and number of sessions etc) and medication delivery (instructions, actual delivery process etc).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No